CLINICAL TRIAL: NCT02173002
Title: Integrated Care for Inflammatory Bowel Disease Patients in the Netherlands With the Novel Telemedicine Tool myIBDcoach: a Randomized Controlled Trial
Acronym: myIBDcoach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: myIBDcoach
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2016-09

CONDITIONS: Inflammatory Bowel Disease
Keywords: Telemedicine; Patient empowerment; Integrated care
MeSH Terms: conditions — Inflammatory Bowel Diseases; Patient Participation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): Standard care
  Interventions: Other: Standard care
- myIBDcoach (Experimental): myIBDcoach
  Interventions: Other: myIBDcoach

INTERVENTIONS:
Other: myIBDcoach
  Arms: myIBDcoach
Other: Standard care
  Arms: Standard care

SUMMARY:
Inflammatory bowel diseases (IBD) is an invalidating disease mainly diagnosed in young people. The disease is characterized by a heterogenic phenotype and the disease course by flares and remissions. As in most chronic diseases the economic burden of IBD is important due to direct health care costs and disability. Health care reorganization for IBD patients in the Netherlands is necessary for several reasons. First chronic (sub)clinical mucosal inflammation results in irreversible bowel damage and complications and none of the presently available drugs is effective for all patients and many drugs have possible severe side effects. To prevent complications of the disease and side effects IBD should be monitored carefully. In the Netherlands however there is a shortage of gastroenterologists where the incidence of IBD is rising. Secondly evidence exists that direct involvement of health care workers, patient empowerment and integrated care can improve the outcome of chronic diseases. Thirdly many clinically relevant aspects (e.g. malnutrition) of this complex disease are not systematically followed in routine care. Finally the government demands registration of efficacy endpoints for expensive drugs in the near future. Therefore the investigators developed a web-based Telemedicine tool for IBD patients in collaboration with the Dutch IBD patient's organization (CCUVN). "myIBcoach" contains E-learning modules, monitors disease activity, disability, quality of life, adherence, infections, smoking status, side effects, stress and malnutrition on fixed time points with validated questionnaires, allows the patient to communicate with health care workers and gives feedback to the back office and the patient. A feasibility study in 30 IBD patients in 3 centres showed a high satisfaction and compliance of IBD-patients and health care workers with this telemedicine tool.

The aim of this study is to compare standard care for IBD patients in 3 hospitals with a care via the telemedicine tool myIBDcoach.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed IBD
* Age 18-75 years
* Patients who have access to internet by computer, tabloid or smartphone

Exclusion Criteria:

* Not able to give informed consent
* Not able to understand and use the Dutch language
* In the two weeks after a hospital admission patients can not be included

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Outpatient hospital visits | 1 year
  Amount of outpatient hospital visits between the two study-arms
Satisfaction | 1 year
  Questionnaire: Patient reported satisfaction with IBD care 0-10

SECONDARY OUTCOMES:
Complications (hospital admissions) | 1 year
  Hospital admission rate
Compliance with IBD care | 1 year
Quality of care | 1 year
  Questionnaire: patient reported quality of care 0-10
Disease specific knowledge | 1 year
  Questionnaire: How do you score your IBD specific knowledge on a scale from 0-10?
Knowledge about treatment | 1 Year
  Questionnaire: How do you score your knowledge about the medication you use on a scale from 0-10?
Medication Adherence | 1 year
  Morisky Medication Adherence Scale
Quality of life | 1 year
  Short IBD questionnaire EQ-6D
Disease activity | 1 year
  Monitor IBD At Home score
Smoking | 1 year
  Change of smoking habits after 1 year
Health care consumption | 1 year
  Questionnaire every 3 months
Self-efficacy | 1 year
  IBD self-efficacy scale

CONTACTS AND LOCATIONS:
Overall Officials: M. Pierik, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] de Jong MJ, Boonen A, van der Meulen-de Jong AE, Romberg-Camps MJ, van Bodegraven AA, Mahmmod N, Markus T, Dijkstra G, Winkens B, van Tubergen A, Masclee A, Jonkers DM, Pierik MJ. Cost-effectiveness of Telemedicine-directed Specialized vs Standard Care for Patients With Inflammatory Bowel Diseases in a Randomized Trial. Clin Gastroenterol Hepatol. 2020 Jul;18(8):1744-1752. doi: 10.1016/j.cgh.2020.04.038. Epub 2020 Apr 23. PMID 32335133
- [Derived] de Jong MJ, van der Meulen-de Jong AE, Romberg-Camps MJ, Becx MC, Maljaars JP, Cilissen M, van Bodegraven AA, Mahmmod N, Markus T, Hameeteman WM, Dijkstra G, Masclee AA, Boonen A, Winkens B, van Tubergen A, Jonkers DM, Pierik MJ. Telemedicine for management of inflammatory bowel disease (myIBDcoach): a pragmatic, multicentre, randomised controlled trial. Lancet. 2017 Sep 2;390(10098):959-968. doi: 10.1016/S0140-6736(17)31327-2. Epub 2017 Jul 14. PMID 28716313